CLINICAL TRIAL: NCT05328570
Title: Effects of Exercise Training on the Structure and Metabolic Function of Fat Tissue
Brief Title: Comparing the Effects of Exercise on the Structure and Function of Fat Tissue
Acronym: CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Professor of Movement Science and Director of the Substrate Metabolism Laboratory (SML) at the University of Michigan School of Kinesiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00179332
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Adiposity
MeSH Terms: conditions — Obesity | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral Glucose Tolerance Test (Experimental): Subjects will complete an Oral Glucose Tolerance Test in which glucose is given and blood samples are taken every 15 minutes over a 2 hour period to determine how quickly the glucose is cleared from the blood.
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test

INTERVENTIONS:
Diagnostic Test: Oral Glucose Tolerance Test — Subjects will complete an Oral Glucose Tolerance Test in which glucose is given and blood samples are taken every 15 minutes over a 2 hour period to determine how quickly the glucose is cleared from the blood.

SUMMARY:
Assess differences in structure and biological function of abdominal subcutaneous adipose tissue samples collected from adults who exercise regularly vs. a well-matched cohort of non-exercisers.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40 years old
* Body Mass Index: 23-35 kg/m2
* Women must have regularly occurring menses and must be premenopausal

Exclusion Criteria:

* Evidence/history of cardiovascular or metabolic disease
* Medications known to affect lipid or glucose metabolism, or inflammation
* Weight instability ≥ ± 6 pounds in the last 6 months
* Tobacco or e-cigarette users
* Women must not be pregnant or actively lactating
* Blood pressure > 140/90 mmHg

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Blood Glucose Level | 2 hours at Experimental Trial
  mg/dL
Adipose tissue fibrosis | baseline
  Pico-sirius Red stain (percent stained)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Horowitz, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No